CLINICAL TRIAL: NCT00904982
Title: Randomized Trial of Interventions to Improve Warfarin Adherence
Acronym: WIN3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 809166
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-01

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Dilated Cardiomyopathies
Keywords: warfarin; coumadin; adherence; mechanical heart valves
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 Usual Care Group/Control (Other): Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication. The MM can display messages to the participant and can confirm when medication is taken correctly.
  Interventions: Behavioral: Financial Incentive and Med-eMonitor
- 2Med-eMonitor/Reminder (Experimental): Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication and will be set on active mode for this group. The MM will display messages of encouragement to participants and education on the importance of taking their warfarin medication. The Med-eMonitor also features an alarm that will sound to remind participants to take their medication as scheduled.
  Interventions: Device: 2Med-eMonitor
- 3 Incentive Group/Lottery (Experimental): Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication. The MM can display messages to the participant. This group will also be entered into a daily lottery in which he/she can win money. On any given study day, participants have a 1 in 10 chance of winning $10 and 1 in 100 chance of winning $100 when taking their warfarin as prescribed. Participants must take their dose correctly in order to be eligible for the daily lottery.
  Interventions: Behavioral: Financial Incentive and Med-eMonitor
- 4 Combined Group/Lottery and Reminder (Experimental): Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication and will be set on active mode for this group. The MM will display messages of encouragement to participants and education on the importance of taking their warfarin medication. The Med-eMonitor also features an alarm that will sound to remind participants to take their medication as scheduled. Participants in this group will also be entered into a daily lottery. On any given study day, participants have a 1 in 10 chance of winning $10 and 1 in 100 chance of winning $100 when taking their warfarin medication as prescribed. Participants must take their dose correctly in order to be eligible for the daily lottery.
  Interventions: Behavioral: Financial Incentive and Med-eMonitor

INTERVENTIONS:
Behavioral: Financial Incentive and Med-eMonitor — Financial Incentives: Study participants are entered into a daily lottery. It includes a chance to win either $10 or $100 on any given day throughout the participant's duration in the study (6 months). Participants are assigned a number and each day a computer randomly draws a winning number. Participants whose number is drawn can only collect money if they have taken the medication correctly.
  Med-eMonitor: The Med-eMonitor is a device used to measure medication compliance. The device has 5 drawers in which the participants' medication is placed. When a drawer opens, a message displays on the monitor, and asks the participant if he/she is taking his/her medication for the day. The device registers their answers and sends the compliance information via the participants' telephone line nightly to a central study server.
  Arms: 1 Usual Care Group/Control; 3 Incentive Group/Lottery; 4 Combined Group/Lottery and Reminder
Device: 2Med-eMonitor — Med-eMonitor is a device that subjects will be given that will monitor an individual's warfarin adherence.
  Arms: 2Med-eMonitor/Reminder

SUMMARY:
The purpose of this research study is to see if a lottery which provides the opportunity to win money, a reminder system using a "Med-eMonitor", or the combination of both might be useful in helping patients to achieve better control of their anticoagulation therapy. Selection for the arms of the study is randomized by the study computer. Some will participate in the daily lottery only, some with the reminder system only, some with the reminder system and the daily lottery, and some with neither the lottery nor the reminder system.

DETAILED DESCRIPTION:
Eligible subjects will be enrolled in one of the 4 arms of the RCT and followed for 6 months, with the primary outcome of out-of-range INRs. Subjects will be given a Med-eMonitor to connect to their home phone line. For all subjects, these will be used to measure daily adherence. Subjects in the incentive group will be eligible for a daily lottery prize only if, prior to the lottery being resolved, their adherence device has registered adherence to their prescribed warfarin regimen. Subjects in the MM group will have the reminder/feedback features of the Med-eMonitor turned on to provide reminders to take their warfarin as prescribed and standardized messages that will be used to provide feedback in response to their adherence. Subjects in the combined group will be exposed to both the lottery and the activated Med-eMonitor. This trial is a randomized controlled trial.

Both men and women who are at least 18 years of age and have been prescribed anticoagulation medication are eligible to participate.

ELIGIBILITY:
Key Inclusion Criteria

The study population will include all patients at the study sites who:

1. are in the maintenance phase of their warfarin treatment (defined using the standard method as the period of time following 2 consecutive visits, at least 7 days apart, of stable target INR after initiation of the drug)
2. whose providers indicate are expected to stay on treatment for at least 6 months
3. have a target INR of 2 to 3.5
4. had at least one INR out of the participant's target range within 90 days prior to enrollment (excluding the baseline visit) and/or INR at the baseline visit was below the participant's target range
5. have a working analog telephone line.

Of note, patients do not have to be within their target INR range to enroll; we specifically want to include those who are below the target range at the time of study entry because they may be the patients most likely to be non-adherent.

Key Exclusion Criteria Patients will be excluded if they do not meet the above inclusion criteria,

1. have an INR at screening above the target range
2. are less than 18 years of age and cannot or will not give consent
3. cannot read above a 6th grade reading level
4. are enrolled in a clinical trial of warfarin therapy
5. are unable to adequately follow study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, M.D., Ph.D., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania Anticoagulation Management Center, Philadelphia, Pennsylvania
  - Philadelphia Veteran Affairs Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Kimmel SE, Troxel AB, French B, Loewenstein G, Doshi JA, Hecht TE, Laskin M, Brensinger CM, Meussner C, Volpp K. A randomized trial of lottery-based incentives and reminders to improve warfarin adherence: the Warfarin Incentives (WIN2) Trial. Pharmacoepidemiol Drug Saf. 2016 Nov;25(11):1219-1227. doi: 10.1002/pds.4094. Epub 2016 Sep 4. PMID 27592594
- [Derived] Kimmel SE, Troxel AB, Loewenstein G, Brensinger CM, Jaskowiak J, Doshi JA, Laskin M, Volpp K. Randomized trial of lottery-based incentives to improve warfarin adherence. Am Heart J. 2012 Aug;164(2):268-74. doi: 10.1016/j.ahj.2012.05.005. PMID 22877814

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Usual Care Group/Control: Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication. The MM can display messages to the participant and can confirm when medication is taken correctly.
  Financial Incentive and Med-eMonitor: Financial Incentives: Study participants are entered into a daily lottery. It includes a chance to win either $10 or $100 on any given day throughout the participant's duration in the study (6 months). Participants are assigned a number and each day a computer randomly draws a winning number. Participants whose number is drawn can only collect money if they have taken the medication correctly.
  Med-eMonitor: The Med-eMonitor is a device used to measure medication compliance. The device has 5 drawers in which the participants' medication is placed. When a drawer opens, a message displays on the monitor, and asks the participant if he/she
- 3 Incentive Group/Lottery: Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication. The MM can display messages to the participant. This group will also be entered into a daily lottery in which he/she can win money. On any given study day, participants have a 1 in 10 chance of winning $10 and 1 in 100 chance of winning $100 when taking their warfarin as prescribed. Participants must take their dose correctly in order to be eligible for the daily lottery.
  Financial Incentive and Med-eMonitor: Financial Incentives: Study participants are entered into a daily lottery. It includes a chance to win either $10 or $100 on any given day throughout the participant's duration in the study (6 months). Participants are assigned a number and each day a computer randomly draws a winning number. Participants whose number is drawn can only collect money if they have taken
- 4 Combined Group/Lottery and Reminder: Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication and will be set on active mode for this group. The MM will display messages of encouragement to participants and education on the importance of taking their warfarin medication. The Med-eMonitor also features an alarm that will sound to remind participants to take their medication as scheduled. Participants in this group will also be entered into a daily lottery. On any given study day, participants have a 1 in 10 chance of winning $10 and 1 in 100 chance of winning $100 when taking their warfarin medication as prescribed. Participants must take their dose correctly in order to be eligible for the daily lottery.
  Financial Incentive and Med-eMonitor: Financial Incentives: Study participants are entered into a daily lottery. It includes a chance to win either $10 or $100 on an
Period: Overall Study
Arm/Group | 1 Usual Care Group/Control | 2Med-eMonitor/Reminder | 3 Incentive Group/Lottery | 4 Combined Group/Lottery and Reminder
Started | 68 | 67 | 67 | 68
Completed | 66 | 67 | 67 | 68
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 Usual Care Group/Control: Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication. The MM can display messages to the participant and can confirm when medication is taken correctly.Financial Incentive and Med-eMonitor: Financial Incentives: Study participants are entered into a daily lottery. It includes a chance to win either $10 or $100 on any given day throughout the participant's duration in the study (6 months). Participants are assigned a number and each day a computer randomly draws a winning number. Participants whose number is drawn can only collect money if they have taken the medication correctly.
  Med-eMonitor: The Med-eMonitor is a device used to measure medication compliance. The device has 5 drawers in which the participants' medication is placed. When a drawer opens, a message displays on the monitor, and asks the participant if he/she
- 3 Incentive Group/Lottery: Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication. The MM can display messages to the participant. This group will also be entered into a daily lottery in which he/she can win money. On any given study day, participants have a 1 in 10 chance of winning $10 and 1 in 100 chance of winning $100 when taking their warfarin as prescribed. Participants must take their dose correctly in order to be eligible for the daily lottery.Financial Incentive and Med-eMonitor: Financial Incentives: Study participants are entered into a daily lottery. It includes a chance to win either $10 or $100 on any given day throughout the participant's duration in the study (6 months). Participants are assigned a number and each day a computer randomly draws a winning number. Participants whose number is drawn can only collect money if they have taken
- 4 Combined Group/Lottery and Reminder: Participants in this study arm will be given an electronic medication monitoring system called a Med-eMonitor(MM) to use at home. This machine will measure the participant's adherence to taking their medication and will be set on active mode for this group. The MM will display messages of encouragement to participants and education on the importance of taking their warfarin medication. The Med-eMonitor also features an alarm that will sound to remind participants to take their medication as scheduled. Participants in this group will also be entered into a daily lottery. On any given study day, participants have a 1 in 10 chance of winning $10 and 1 in 100 chance of winning $100 when taking their warfarin medication as prescribed. Participants must take their dose correctly in order to be eligible for the daily lottery.Financial Incentive and Med-eMonitor: Financial Incentives: Study participants are entered into a daily lottery. It includes a chance to win either $10 or $100 on an
- Total: Total of all reporting groups
Arm/Group | 1 Usual Care Group/Control | 2Med-eMonitor/Reminder | 3 Incentive Group/Lottery | 4 Combined Group/Lottery and Reminder | Total
Number analyzed (Participants) | 68 | 67 | 67 | 68 | 270
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [60.0 to 71.0] | 62 [55.0 to 67.0] | 62 [51.0 to 68.0] | 61.5 [51.5 to 68.5] | 62 [54 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 21 | 25 | 86
  Male | 45 | 50 | 46 | 43 | 184
Region of Enrollment [Number; unit: participants]
  United States | 68 | 67 | 67 | 68 | 270

OUTCOME MEASURES:

1. Primary Outcome: Improved Warfarin Adherence/% Timeout of Target INR Range
Time Frame: six months
Population: This analysis required multiple INR results. If those were not available for a subject, they were excluded from the primary analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of out of target INR range
Arm/Group | 1 Usual Care Group/Control | 2Med-eMonitor/Reminder | 3 Incentive Group/Lottery | 4 Combined Group/Lottery and Reminder
Number analyzed (Participants) | 66 | 64 | 64 | 67
percentage of out of target INR range | 31.6 [11.1 to 50.5] | 23.8 [8.8 to 36.6] | 30.1 [12.4 to 46.3] | 23.9 [9.9 to 42.7]

ADVERSE EVENTS:
Arm/Group | 1 Usual Care Group/Control | 2Med-eMonitor/Reminder | 3 Incentive Group/Lottery | 4 Combined Group/Lottery and Reminder
Serious Adverse Events (participants affected / at risk) | 4/65 | 4/63 | 4/65 | 5/66
Other Adverse Events (participants affected / at risk) | 1/65 | 3/63 | 2/65 | 5/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Usual Care Group/Control (N=65) | 2Med-eMonitor/Reminder (N=63) | 3 Incentive Group/Lottery (N=65) | 4 Combined Group/Lottery and Reminder (N=66)
Stroke/TIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-CNS Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Major Bleeding (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 2 (2) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Usual Care Group/Control (N=65) | 2Med-eMonitor/Reminder (N=63) | 3 Incentive Group/Lottery (N=65) | 4 Combined Group/Lottery and Reminder (N=66)
Non-Serious Bleeding (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Non-serious Clotting (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No